CLINICAL TRIAL: NCT03528707
Title: Effect of Probiotic Co-administration With Omega-3 Fatty Acids on NAFLD: Randomized Clinical Studies
Brief Title: Effect of Probiotic Co-administration With Omega-3 Fatty Acids on NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Nazarii Kobyliak, Associate Professor of Endocrinology Department, PhD, Bogomolets National Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDO-2
Record Dates: First submitted 2018-05-01; First posted 2018-05-18 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Type2 Diabetes; NAFLD; Probiotic; Omega-3 Fatty Acids
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization was done by the study statistician based on a computer-generated list. The groups were homogeneous according to age, sex and diagnostic criteria. The assignment of groups was blind to participants, research staff and outcome assessors moreover, to maintain blind parallel study the statistician was not aware of the allocation of participants to intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic-omega (Active Comparator): Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) of gel per day.
  Interventions: Dietary Supplement: Symbiter-Omega
- placebo (Placebo Comparator): Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) of gel per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Symbiter-Omega — "Symbiter Omega" which contains combination of flax and wheat germ oil (250 mg of each, concentration of omega-3 fatty acids 1-5%), supplemented with biomass of 14 alive probiotic strains: Lactobacillus + Lactococcus (6×1010 CFU/g), Bifidobacterium (1×101
  Arms: probiotic-omega
Dietary Supplement: Placebo — Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) of gel per day
  Arms: placebo

SUMMARY:
One of the potential ideal strategy for NAFLD treatment may be manipulation with gut microbiota. Probiotics are defined as live microorganisms that, when administered in adequate amounts, confer a health benefit on the host. Omega-3 fatty acids belong to the family of polyunsaturated fatty acids. They are known to exert a strong positive influence on metabolism and inflammation. The data from animal studies suggested that both probiotics and omega-3 can affect body weight, influence on glucose and fat metabolism, improve insulin sensitivity and reduce chronic systemic inflammation. In respect to experimental data, the current study aim was to provide double-blind single center RCT, for study the efficacy of co-administration of probiotic with omega-3 vs. placebo in type 2 diabetes patient with NAFLD detected on ultrasonography

DETAILED DESCRIPTION:
In this single-center double-blind, placebo controlled, parallel group study, 48 type 2 diabetes patients from the Kyiv City Clinical Endocrinology Center were selected. They were randomly assigned to receive "Symbiter Omega" or placebo for 8 weeks, administered as a sachet formulation in double-blind treatment. Randomization was done by the study statistician based on a computer-generated list. The groups were homogeneous according to age, sex and diagnostic criteria. The assignment of groups was blind to participants, research staff and outcome assessors moreover, to maintain blind parallel study the statistician was not aware of the allocation of participants to intervention.

The "Symbiter Omega" was supplied by Scientific and Production Company "O.D. Prolisok". It contains combination of flax and wheat germ oil (250 mg of each, concentration of omega-3 fatty acids 1-5%), supplemented with biomass of 14 alive probiotic strains: Lactobacillus + Lactococcus (6×1010 CFU/g), Bifidobacterium (1×1010/g), Propionibacterium (3×1010/g), Acetobacter (1×106/g) genera. Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) of probiotic-omega and placebo per day. All sachets were identical with similar organoleptic characteristics (e.g., taste and appearance).

The pre-randomization period was designed to minimize the effects of dietary changes on metabolic markers. For this purpose, 2 weeks before the study start, after inform consent signed, patients were instructed in one-on-one sessions with a dietitian to follow a therapeutic lifestyle-change diet as classiﬁed by the NCEP. In addition, participants were instructed to continue with stable anti-hyperglycemic treatment and received standardized mild physical training for 1 hour per day.

Patients who underwent the study were instructed to take the trial medication as prescribed. Throughout the study, weekly phone follow-up visits were provided for assessment of compliance, adherence to the protocol, as well as the recording of adverse events. The effectiveness of therapy was compared and evaluated separately in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* adult participants (ages 18-75, BMI ≥25 kg/m2) diagnosed with NAFLD according to the recommendations of the American Gastroenterology Association (AGA) and American Association for the Study of Liver Disease (AASLD);
* the diagnosis of fatty liver was based on the results of abdominal ultrasonography. Of 4 known criteria (hepato-renal echo contrast, liver brightness, deep attenuation, and vascular blurring), the participants were required to have hepato-renal contrast and liver brightness to be given a diagnosis of NAFLD.
* type 2 diabetes treated with diet and exercise alone or metformin, SUs and insulin at stable dose at least 4 weeks prior to the commencement of the study;
* AST and ALT ≤3x upper limit of normal.

Exclusion Criteria:

* alcohol abuse (>20 g/day (2 standard drinks) in women or > 30 g/d (3 drinks) in men over a two-year period);
* chronic viral hepatitis (associated with HBV, HCV, HDV infection);
* drug-induced liver disease, Wilson's disease, hereditary deficiency of antitrypsin-1 and idiopathic hemochromatosis;
* history of decompensated liver disease including ascites, encephalopathy or variceal bleeding;
* regular use of a probiotic or prebiotic supplement within 3 months prior to enrollment;
* antibiotic use within 3 months prior to enrollment;
* uncontrolled cardiovascular or respiratory disease, active malignancy, or chronic infections;
* use of agents such as vitamin E, omega-3 fatty acids or medications with evidence for effects on NAFLD (pioglitazone, GLP-1 analogues, dipeptidyl peptidase IV inhibitors, ursodeoxycholic acid);
* and presence of active infection, pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2015-12-22 (Actual); Study Completion 2016-01-28 (Actual)

PRIMARY OUTCOMES:
fatty liver index (FLI) | 8 weeks compared to baseline
  FLI = [e 0.953*loge (triglycerides) + 0.139*BMI + 0.718*loge (ggt) + 0.053*waist circumference - 15.745) / (1 + e 0.953*loge (triglycerides) + 0.139*BMI + 0.718*loge (ggt) + 0.053*waist circumference - 15.745)] × 100
liver stiffness (LS) | 8 weeks compared to baseline
  liver stiffness (LS) was measured by Shear Wave Elastography (SWE) and expressed in kPa.

SECONDARY OUTCOMES:
ALT | 8 weeks compared to baseline
  ALT in IU/L
AST | 8 weeks compared to baseline
  AST in IU/L
γ-GT | 8 weeks compared to baseline
  γ-GT in IU/L
Total Cholesterol (TC) | 8 weeks compared to baseline
  TC in mmol/l
Tryglicerides (TG) | 8 weeks compared to baseline
  TG in mmol/l
LDL-Cholesterol (LDL-C) | 8 weeks compared to baseline
  LDL-C in mmol/l
VLDL-Cholesterol (VLDL-C) | 8 weeks compared to baseline
  VLDL-C in mmol/l
HDL-Cholesterol (HDL-C) | 8 weeks compared to baseline
  HDL-C in mmol/l
cytokines levels | 8 weeks compared to baseline
  TNF-α, IL-1β, IL-6, IL-8, INF-γ in pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Galyna Mykhalchyshyn, PhD, Principal Investigator — Bogomolets National Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kobyliak N, Abenavoli L, Falalyeyeva T, Mykhalchyshyn G, Boccuto L, Kononenko L, Kyriienko D, Komisarenko I, Dynnyk O. Beneficial effects of probiotic combination with omega-3 fatty acids in NAFLD: a randomized clinical study. Minerva Med. 2018 Dec;109(6):418-428. doi: 10.23736/S0026-4806.18.05845-7. Epub 2018 Sep 13. PMID 30221912